CLINICAL TRIAL: NCT05331989
Title: Smartphone Addiction and Temporomandibular Joint Dysfunction in Individuals With Nonspecific Neck Pain
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ayşe Abit Kocaman, Principal Investigator, Kırıkkale University
Other Study IDs: SmartphoneAddictionandneckpain
Record Dates: First submitted 2022-04-10; First posted 2022-04-18 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Smartphone Addiction, Temporomandibular Joint Dysfunction
MeSH Terms: conditions — Internet Addiction Disorder; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient group,healthy group: Cranio- Cervical Flexion Test, cervical mobility, Pressure Pain Threshold,Functional evaluation of the temporomandibular joint,Pittsburg Sleep Quality Index
  Interventions: Other: patient group/ healthy group

INTERVENTIONS:
Other: patient group/ healthy group — Cranio- Cervical Flexion Test, cervical mobility, Pressure Pain Threshold,Functional evaluation of the temporomandibular joint,Pittsburg Sleep Quality Index

SUMMARY:
It has been reported that excessive use of smartphones increases the stress on the cervical spine, and changes in cervical curvature and pain in the muscles around the neck are associated with the increase in stress. Studies have reported that smartphone users with addictions have neck pain (68%), upper back pain (62%), right shoulder pain (52%), left shoulder pain (46%), and right hand pain (46%). As a result of our study, the frequency of smartphone addiction and temporomandibular joint dysfunction and related factors in individuals with nonspecific neck pain were examined and the results we obtained will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Presence of neck pain lasting at least 6 months
* Being between the ages of 18-45
* Individuals with a score between 10-40 points according to the Neck Disability Index
* Individuals who have never had a history of shoulder or neck surgery

Exclusion Criteria:

* Individuals with signs of radicular pain (positive neck distraction test, Spurling's neck compression test, and Adson's test)
* Individuals who get less than 10 points or more than 40 points according to the Neck Disability Index
* Those with a previous history of shoulder and neck surgery
* Individuals with accompanying shoulder pain
* Individuals with spinal cord tumors
* Individuals with meningeal tumors
* Individuals who do not want to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with nonspecific neck pain, individuals who voluntarily agreed to participate in our study and signed the consent form
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Cranio- Cervical Flexion Test | Day 1
  An inflatable pressure unit (StabilizerTM, Chattanooga Group, Inc., Hixson, TN) will be used during testing.
Evaluation of cervical mobility | Day 1
  Cervical region flexion, extension, lateral flexion and rotation movements will be evaluated with Baseline Bubble Inclinometer.
Evaluation of Pressure Pain Threshold | Day 1
  Pressure pain threshold assessment will be performed with an algometer, which is an objective assessment method.Measurements will be made from three different regions: anterior temporal muscle body, masseter muscle body and TMJ (lateral to the mandibular condyle).
Functional evaluation of the temporomandibular joint | Day 1
  The Helkimo Clinic Craniomandibular Index will be used in the evaluation of TMJ (5). This index consists of 5 subsections: pain on muscle palpation, pain on TMJ palpation, pain on mandible functions, TMJ functions (sound, gliding at maximum opening, luxation and/or locking) and mandible movement capacity.
Smartphone Addiction Scale Short Form | Day 1
  Each item is scored between 1-6. The high score informs about the severity of smartphone addiction. Those who have a total score above 29.50 are considered as smartphone addiction.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Day 1
  It is a reliable, valid and standardized scale that measures sleep quality over a one-month period and provides clinical evaluation of various sleep disorders that may affect sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Abit Kocaman, PhD, Principal Investigator — Kırıkkale University
Locations (1):
- Ayşe Abit Kocaman, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Can HB, Tuna F. Relation between endurance of deep cervical flexor muscles and physical activity level, perceived stress, sleep quality, and smartphone addiction. Cranio. 2022 Mar;40(2):126-134. doi: 10.1080/08869634.2020.1724457. Epub 2020 Feb 6. PMID 32028877